CLINICAL TRIAL: NCT03224312
Title: Chongqing Primary Aldosteronism Study
Status: Recruiting | Type: Observational
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Qifu Li, Director of endocrinology, First Affiliated Hospital of Chongqing Medical University
Other Study IDs: CONPASS
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Primary Aldosteronism
Keywords: Primary aldosteronism; cardiovascular events; cerebrovascular events
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma and complete blood cell, adrenals.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary aldosteronism: screened, confirmed and subtyped according to the guidelines.
  Interventions: Other: no intervention
- Essential hypertension: screened for PA and excluded the diagnosis of PA as well as other secondary hypertesion
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
We intends to conduct a series of original clinical research about PA, and establish a large cohort of PA and essential hypertension patients with long-term follow-up of cardiovascular events, renal end points etc. We will establish a large sample of blood, urine, adrenal tissue of the subjects, and the genomics,metabonomics, proteomics database, to explore the mechanism of the PA and target organ damage, risk factors, diagnostic methods and biomarkers.

DETAILED DESCRIPTION:
This study will include the subjects of a series of studies on hypertension conducted by our team, including essential hypertension, PA subjects, and establish a large sample database and specimen bank through follow-up and omics analysis.

ELIGIBILITY:
Inclusion Criteria:

1. hypertensive patients who completed ARR screening and necessary further tests;
2. Voluntary to sign the informed consent.

Exclusion Criteria:

1. patients with severe cardiac, hepatic or renal dysfunction;
2. suspicious or confirmed other types of secondary hypertension, including Cushing's syndrome, pheochromocytoma and renal artery stenosis et al.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hypertensive patients who completed ARR screening and necessary further tests and Voluntary to be followed up will be included.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
numbers of patients who develop cardiovascular events | 1-15 years
  compare the long-term cardiovascular and cerebrovascular events in patients with primary aldosteronism and essential hypertension

SECONDARY OUTCOMES:
estimated glomerular filtration rate (eGFR) | 1-15 years
  Compare the incidence of hypertensive nephropathy between two groups (based on eGFR)
The incidence of new atrial fibrillation | 1-15 years
  Compare the occurrence of new atrial fibrillation between patients with primary aldosteronism and essential hypertension
The incidence of left ventricular hypertrophy | 1-15 years
  Compare the occurrence of left ventricular hypertrophy between patients with primary aldosteronism and essential hypertension
the variation of carotid intima-media thickness | 1-15 years
  Compare the occurrence of the variation of carotid intima-media thickness between patients with primary aldosteronism and essential hypertension
subgroup analysis of cardiovascular events | 1-15 years
  Compare the cardiovascular and cerebrovascular risk between unilateral PA and idiopathic bilateral adrenal hyperplasia
quality of life score | 1-15 years
  Compare the quality of life between unilateral PA and idiopathic bilateral adrenal hyperplasia by the questionnaire.
Cardiovascular risk score | 1-15 years
  To investigate what kind of cardiovascular risk score can better predict cardiovascular risk of PA

CONTACTS AND LOCATIONS:
Overall Officials: Qifu Li, phD, Study Chair — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- Qifu Li, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Background] Williams TA, Lenders JWM, Mulatero P, Burrello J, Rottenkolber M, Adolf C, Satoh F, Amar L, Quinkler M, Deinum J, Beuschlein F, Kitamoto KK, Pham U, Morimoto R, Umakoshi H, Prejbisz A, Kocjan T, Naruse M, Stowasser M, Nishikawa T, Young WF Jr, Gomez-Sanchez CE, Funder JW, Reincke M; Primary Aldosteronism Surgery Outcome (PASO) investigators. Outcomes after adrenalectomy for unilateral primary aldosteronism: an international consensus on outcome measures and analysis of remission rates in an international cohort. Lancet Diabetes Endocrinol. 2017 Sep;5(9):689-699. doi: 10.1016/S2213-8587(17)30135-3. Epub 2017 May 30. PMID 28576687
- [Background] Monticone S, Burrello J, Tizzani D, Bertello C, Viola A, Buffolo F, Gabetti L, Mengozzi G, Williams TA, Rabbia F, Veglio F, Mulatero P. Prevalence and Clinical Manifestations of Primary Aldosteronism Encountered in Primary Care Practice. J Am Coll Cardiol. 2017 Apr 11;69(14):1811-1820. doi: 10.1016/j.jacc.2017.01.052. PMID 28385310
- [Background] Stowasser M, Gordon RD. Primary Aldosteronism: Changing Definitions and New Concepts of Physiology and Pathophysiology Both Inside and Outside the Kidney. Physiol Rev. 2016 Oct;96(4):1327-84. doi: 10.1152/physrev.00026.2015. PMID 27535640
- [Derived] He C, Li R, Yang J, Shen H, Wang Y, Chen X, Luo W, Zeng Q, Ma L, Song Y, Cheng Q, Wang Z, Wu FF, Li Q, Yang S, Hu J. Optimizing the aldosterone-to-renin ratio cut-off for screening primary aldosteronism based on cardiovascular risk: a collaborative study. Clin Exp Hypertens. 2024 Dec 31;46(1):2301571. doi: 10.1080/10641963.2023.2301571. Epub 2024 Jan 25. PMID 38270079
- [Derived] Yang Y, Williams TA, Song Y, Yang S, He W, Wang K, Cheng Q, Ma L, Luo T, Yang J, Reincke M, Burrello J, Li Q, Mulatero P, Hu J. Nomogram-Based Preoperative Score for Predicting Clinical Outcome in Unilateral Primary Aldosteronism. J Clin Endocrinol Metab. 2020 Dec 1;105(12):dgaa634. doi: 10.1210/clinem/dgaa634. PMID 32898224
- [Derived] Wang K, Hu J, Yang J, Song Y, Fuller PJ, Hashimura H, He W, Feng Z, Cheng Q, Du Z, Wang Z, Ma L, Yang S, Li Q. Development and Validation of Criteria for Sparing Confirmatory Tests in Diagnosing Primary Aldosteronism. J Clin Endocrinol Metab. 2020 Jul 1;105(7):dgaa282. doi: 10.1210/clinem/dgaa282. PMID 32449927